CLINICAL TRIAL: NCT03301974
Title: A Comparison Between Surgical Techniques for Securing Conjunctival Autografting in Primary Pterygium Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Fathy Ahmed Oraby, Specialist of ophthalmology, El-Mabarah hospital for Health insurance, Assuit, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17200138
Record Dates: First submitted 2017-09-27; First posted 2017-10-04 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conjunctival autograft with fibrin glue (Experimental): Conjunctival autograft with fibrin glue done for patients of group 1 after pterygium excision
  Interventions: Procedure: conjunctival autograft with fibrin glue
- sutured conjunctival autograft (Experimental): Sutured conjunctival autograft done for patients of group 2 after pterygium excision
  Interventions: Procedure: sutured conjunctival autograft
- sutureless and glue-free conjunctival autograft (Experimental): Sutureless, glue-free conjunctival autograft done for patients of group 3 after pterygium excision
  Interventions: Procedure: sutureless and glue-free conjunctival autograft

INTERVENTIONS:
Procedure: conjunctival autograft with fibrin glue — Simple pterygium excision under local anesthesia performed then closure of the bare sclera by fibrin glued conjunctival autograft in 20 eyes of 20 patients (group 1).
  Arms: conjunctival autograft with fibrin glue
Procedure: sutured conjunctival autograft — Simple pterygium excision under local anesthesia performed then closure of the bare sclera by sutured conjunctival autograft in 20 eyes of 20 patients (group 2).
  Arms: sutured conjunctival autograft
Procedure: sutureless and glue-free conjunctival autograft — Simple pterygium excision under local anesthesia performed then closure of the bare sclera by sutureless and glue free conjunctival autograft in 20 eyes of 20 patients (group 3)
  Arms: sutureless and glue-free conjunctival autograft

SUMMARY:
Pterygium is a fibrovascular wing shaped encroachment of conjunctival fold on to the cornea with elastotic degeneration of a subconjunctival tissue, The standard treatment for pterygium is surgical excision, but the recurrence rate after surgery can be as high as 24%-89%, which compromises outcomes. Based on the simple excision of pterygium, multiple strategies and techniques have been developed to reduce the high rate of pterygium recurrence. The investigators aim was to compare the safety, efficacy, overall patient satisfaction and recurrence rate of suturing, fibrin gluing and sutureless glue-free technique for attaching conjunctival autograft in primary pterygium surgery.

DETAILED DESCRIPTION:
Design: Prospective randomized comparative interventional clinical study Setting: Assiut university hospital & El-Mabarah hospital for health insurance Methods: The study included 60 eyes of 60 consecutive patients of primary nasal pterygium were enrolled in the study. Simple excision under local anesthesia was performed then closure of the bare sclera by conjunctival autograft with fibrin glue in 20 eyes of 20 patients (group 1), versus sutured free conjunctival autograft in 20 eyes of 20 patients (group 2) ), versus sutureless and glue-free conjunctival autograft in 20 eyes of 20 patients (group 3).

ELIGIBILITY:
Inclusion Criteria:

1. Patients complaining of primary Progressive nasal pterygium.
2. Patients with pterygium threatening the visual axis.

Exclusion Criteria:

1. Double head pterygium.
2. Pseudopterygium
3. Recurrent pterygium
4. Patients with history of any bleeding abnormalities
5. Patients with ocular surface diseases eg- blepharitis, Sjogren syndrome and dry eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-24 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | 6 months postoperatively
  The main postoperative primary outcomes measure the recurrence rate

SECONDARY OUTCOMES:
Graft stability | 1 day, 2 day, 1 week, 1 month 3 months and 6 months postoperatively
  postoperative Graft stability rated from grade 0 to 4 using a 5 point scale
Postoperative inflammation | 1 day, 2 day, 1 week, 1 month 3 months and 6 months postoperatively
  postoperative inflammation rated from grade 0 to 4 using a 5 point scale
Postoperative discomfort | 1 day, 2 day, 1 week, 1 month 3 months and 6 months postoperatively
  postoperative discomfort rated from 0 to 10 on the Visual Analogue Scale (VAS)
Overall patient satisfaction | 1 day, 2 day, 1 week, 1 month 3 months and 6 months postoperatively
  Overall satisfaction with the procedure 4 weeks post-operatively will recorded as four grades 0= unsatisfied, 1= low satisfaction, 2= moderate satisfaction and 3= highly satisfied, the data were collected as mean scores and recorded. The three groups will compared for overall satisfaction.
Complications | 1 day, 2 day, 1 week, 1 month 3 months and 6 months postoperatively
  Complications recorded including, persistent epithelial defect, dellen, inclusion cyst, pyogenic granuloma, conjunctival edema, corneal scleral necrosis, infective scleritis, keratitis and endophthalmitis.